CLINICAL TRIAL: NCT07225595
Title: Supporting Pregnant Patients as They Face a Changing Landscape of Prenatal Genetic Tests and Post-diagnosis Options (Shifting Options)
Brief Title: Shifting Options Study
Status: Active, not recruiting | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 24-826
Record Dates: First submitted 2024-11-19; First posted 2025-11-06 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Prenatal Care; Prenatal Diagnosis
Keywords: shared decision-making; informed decision-making; prenatal screening and diagnostic testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient participants, Group 1 (N=60): Group 1 consists of patient participants. Patient participants will be fit into one of the following sub-categories: (Group 1A, N=20) patients who initiate care in the 1st or 2nd trimester of pregnancy, (Group 1B, N=20) pregnant patients with similar characteristics to category 1, but who have scheduled their 2nd trimester anatomical ultrasound at one of the study sites, and (Group 1C, N=20) patients who are 1-12 months postpartum and delivered at one of the participating sites.
- Clinician participants, Group 2 (N=50): Participants (N=50) include primary OB providers, maternal-fetal specialists, genetic counselors and genetic specialists who provide outpatient obstetric care and practice at one of the outpatient clinics of the study sites.

SUMMARY:
The goal of Shifting Options is to create strategies and resources that will facilitate informed decision-making about prenatal screening and diagnostic testing (PS&D) for all pregnant patients. Shifting Options will determine how rapid changes in PS&D and post-diagnosis options affect the nature and timing of resources and support patients need to make informed PS&D decisions.

To achieve this goal, patient participants will be interviewed to identify their PS&D decision-making needs. Then, clinician participants input will be added on how best to implement strategies that address those needs.

DETAILED DESCRIPTION:
Study overview:

Prenatal genetic screening and diagnostic tests (PS&D) contribute to optimal fetal/neonatal outcomes through the delivery of high-quality prenatal care. While PS&Ds are an important part of prenatal care delivery, advances in PS&D present a challenge to ensure pregnant patients have the information and resources to make informed decisions about their use. This complexity is due to significant advances in prenatal genomics that continue to introduce new PS&D, increasing the number of conditions that can be detected before birth. It is also due to parallel changes in maternal-fetal medicine, pediatrics, and reproductive policy that rapidly change the options available if a fetal genetic condition is diagnosed. Consequently, patients face a growing challenge in making informed decisions about a moving target of testing and post-diagnosis options. As a result, a serious and urgent unmet clinical problem has emerged: There is a lack of evidence-based guidance to support an individualized informed decision-making process for patients amidst an increasingly complex set of reproductive healthcare choices. The objective of our study is to generate strategies and resources that will facilitate informed decision-making about PS&D by diverse populations of pregnant patients. This project is a first step to identifying what strategies may be needed to best prepare patients for this increasingly complex decision-making landscape.

Methods:

The study will engage with two populations: (Group 1) the investigators will conduct in-depth interviews with patients to identify key factors that impact the decision-making and the resources needed to support that process, and (Group 2) with prenatal clinicians to obtain input on patient-reported decision-making priorities and resources to frame a set of initial considerations for strategy and tool implementation. Since this is an observational study, there will be no intervention, neither group will be randomized.

Study Population

Patient participants, Group 1:

Patient participants will be enrolled into 1 of 3 sub-categories: (Group 1A) includes patients who initiate care in the 1st or 2nd trimester of pregnancy to understand decision-making factors as a function of access to prenatal care, (Group 1B) includes pregnant patients with similar characteristics to category 1, but are scheduled their 2nd trimester anatomical ultrasound at one of the study sites, and (Group 1C) includes patients who are 1-12 months postpartum and delivered at one of the participating sites.

Clinician participants, Group 2:

Participants include primary OB providers, maternal-fetal specialists, genetic counselors and genetic specialists who provide outpatient obstetric care and practice at one of the outpatient clinics of the study sites.

Data Collection

Group 1 (qualitative interviews):

After completing an informed consent document, all Group 1 participants will complete an enrollment survey to collect demographic information. A member of the research team will then conduct individual semi-structured interviews with each participant. The interview guide was developed in collaboration with content experts in obstetrics, neonatology, pediatrics, genetics, medical decision-making and ethics. The interview guide will examine participants' informational and decision-making needs with respect to their (1) familiarity with the concepts associated with PS&D, including test characteristics and implications of screens and diagnostic tests, notions of average-risk and increased-risk based on reproductive history or test result, (2) familiarity with current and forthcoming perinatal, neonatal, and pediatric interventions to improve outcomes of a child with a genetic condition or, for those participants who agree to discuss questions about pregnancy termination, familiarity with access to abortion services, (3) preferences regarding the decisional and informational domains needed when considering PS&D use, (4) ways to approach making complex medical decisions, including tolerance of uncertainty and risk and how those preferences may change with gestational age and acquiring in-formation about the fetus, and (5) barriers and facilitators to support an informed decision-making process about initiating PS&D that integrates information about post-diagnosis that align with the patients' needs and goals. Data collection activities will be guided by specific Human Subject Protections to ensure safeguards are in place for participants who elect to discuss opinions or actions related to pregnancy termination. All sessions will be audio-recorded for data analysis purposes.

Group 2 (qualitative interviews):

After completing an informed consent document, all Group 2 participants will complete an enrollment survey to collect demographic information. A member of the research team will then conduct individual semi-structured interviews with each participant. Interviews will be completed using the Implementation Roadmap developed by the ORD Quality Enhancement Research Initiative to guide seeking clinicians' input on patient-reported needs. This roadmap outlines three phases to guide implementation and dissemination of novel interventions. Although given the stage of this work, the investigators will focus on Phases 1 and 2 to identify how patient-reported decision-making needs may be integrated into clinical workflows: Phase 1-Planning, Framing, and Aligning Interested Parties, and Phase 2-Implementation Process Data Collection. The investigators will use the Implementation Planning Assessment Tool (IPA Tool) to develop and structure the interview guide. This will include open-ended questions about how to translate patient-reported needs into approaches that can be effectively integrated into prenatal care delivery. The interview guide will include questions about the proposed Phase 2 implementation plan. Specifically, how the process will be studied, measured, and assessed. The final section of interview guide will contain a set of questions to collect demographic and practice-related information. All sessions will be audio-recorded for data analysis purposes.

Data Analysis:

Audio-recordings will be transcribed verbatim and verified for accuracy. The investigators will use standard qualitative data analysis techniques based on grounded theory for analysis and interpretation of all qualitative data, including decisions regarding theoretical saturation to end data collection. Group 1 themes identified will be contextualized with information about the trimester of pregnancy, gravity/parity, and previous pregnancies. Group 2 themes will consider information about degree type, years in practice, and clinical setting. The investigators will conduct matrix analyses to compare themes and findings across these two groups to identify areas of alignment and discordance with Group 1 resources and Group 2 input on the ability to implement those resources in prenatal care delivery.

ELIGIBILITY:
Group 1 Inclusion Criteria:

1. 18 years of age or older
2. Ability to read and speak English
3. Able to provide consent to participate in the study
4. Have a viable intrauterine pregnancy (IUP) or 1-12 postpartum
5. Offered routine aneuploidy screening and diagnostic testing
6. Seeking care at one of the participating study sites

Group 1 Exclusion Criteria:

1. <18 years of age or older
2. Inability to read and speak English
3. Not able to provide consent to participate in the study
4. Does not have a viable intrauterine pregnancy (IUP) or is not 1-12 postpartum
5. Was not offered routine aneuploidy screening and diagnostic testing
6. Is not seeking care at one of the participating study sites

Group 2 Inclusion Criteria:

1. Board eligible clinicians who provide prenatal care (includes OB/GYNs, CNMs, NPs, MFMs, GC, etc.)
2. Provide outpatient obstetric care
3. Practice at one of the study sites

Group 2 Exclusion Criteria:

1. Not board eligible clinicians who provide prenatal care (includes OB/GYNs, CNMs, NPs, MFMs, GC, etc.)
2. Does not provide outpatient obstetric care
3. Does not practice at one of the study sites

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant or postpartum females
Study Population: Group 1 participants include those who are in their 1st or 2nd trimester of pregnancy or are 1-12 months post partum (Groups 1A, 1B and 1C). These participants will be seeking prenatal or postpartum care at one of the participating study sites.
  Group 2 participants will be practicing and seeing patients at one of the study sites outpatient locations.
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Qualitative analysis completed using Grounded Theory in examining patient participant interviews to uncover emerging codes, memos, and themes that build strategies to support prenatal screening and diagnostic testing informed decision-making. | 12 months
  The study outcome will include qualitative interview data about the prenatal screening and diagnostic testing decision-making process and a foundation for innovative strategies to support patients' informed decision-making with tandem changes in prenatal genomics and available post-diagnosis options. This work will allow researchers to characterize how patients conceptualize the shifting landscape of testing and post-diagnosis options about prenatal screening and diagnostic testing.
Qualitative analysis completed using Grounded Theory in examining provider participant interviews to uncover emerging codes, memos, and themes that build strategies or tools to support prenatal screening and diagnostic testing informed decision-making. | 12 months
  The study outcome will include qualitative interview data about the prenatal screening and diagnostic testing decision-making process and a foundation for innovative strategies to support patients' informed decision-making with tandem changes in prenatal genomics and available post-diagnosis options. This work will allow researchers to characterize how providers can support patients with the shifting landscape of testing and post-diagnosis options about prenatal screening and diagnostic testing and how these resources would best be implemented into prenatal care delivery within the clinical setting.

CONTACTS AND LOCATIONS:
Overall Officials: Ruth M Farrell, MD, MA, Principal Investigator — The Cleveland Clinic
Locations (2):
- United States (2):
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio